CLINICAL TRIAL: NCT01334944
Title: A Multi-Center, Open-Label, Surveillance Trial To Evaluate The Safety and Efficacy of a Shortened Infusion Time of Intravenous Ibuprofen.
Brief Title: Surveillance Trial to Evaluate a Shortened Infusion Time of Intravenous Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL-015
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2016-07

CONDITIONS: Pain; Fever
Keywords: Pain; Fever
MeSH Terms: conditions — Pain; Fever | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous ibuprofen (Experimental): Intravenous ibuprofen (400 mg or 800 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 5-10 minute Treatment Period.
  Interventions: Drug: Intravenous ibuprofen

INTERVENTIONS:
Drug: Intravenous ibuprofen — 400 mg or 800 mg intravenous ibuprofen administered intravenously over 5-10 minutes
  Other Names: Caldolor

SUMMARY:
The primary objective of this study is to determine the safety of a single dose of intravenous ibuprofen administered over 5-10 minutes for the treatment of fever or pain in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Pain: Patients with baseline Visual Analog Scale assessment >3, -and/or- Fever: Patients with temperature >101°F.

Exclusion Criteria:

1. Patients with inadequate IV access
2. Patients <18 years of age
3. History or allergy or hypersensitivity to any component of intravenous ibuprofen, aspirin (or aspirin related products) or non-steroidal anti-inflammatory drug (NSAIDs)
4. Active hemorrhage or clinically significant bleeding
5. Pregnant or nursing
6. Patients in the peri-operative period in the setting of coronary artery bypass graft (CABG) surgery
7. Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions
8. Refusal to provide written authorization for use and disclosure of protected health information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art P Wheeler, M.D., Study Director — Cumberland Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - UCSD, San Diego, California
  - Danbury, Danbury, Connecticut
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Grady, Atlanta, Georgia
  - Beth Israel Deaconnes MC, Boston, Massachusetts
  - Columbia, New York, New York
  - The University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Fairview, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Lankenau, Wynnewood, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients in the hospital setting experiencing pain and/or fever.
Pre-assignment Details: Patients who met all the inclusion and none of the exclusion criteria during the Screening /Baseline Period were enrolled into the study.
  Subjects could not have a history of allergy or hypersensitivity to any component of intravenous ibuprofen, aspirin (or aspirin related products) or NSAIDS.
Groups:
- Fever: Intravenous ibuprofen (400 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 5-10 minute Treatment Period. Patients may receive up to five additional doses of 400 mg (every four hours), as determined by the investigator
- Pain: Intravenous ibuprofen (800 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 5-10 minute Treatment Period. Patients may receive up to three additional doses of 800 mg (every six hours), as determined by the investigator
Period: Overall Study
Arm/Group | Fever | Pain
Started | 11 | 139
Received Singel Dose | 1 | 96
Received Multiple Doses | 10 | 43
Completed | 11 | 139
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous Ibuprofen
Number analyzed (Participants) | 150
Age, Customized [Number; unit: years] — Greater than or equal to 18 years of age
  years
    Greater than or equal to 18 years of age | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 34
  White | 106
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The incidence of treatment-emergent serious adverse events occurring in the six hours following administration of the last dose of intravenous ibuprofen
Time Frame: 6 hours
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
Number of Serious Adverse Events | 0 | 0

2. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The incidence of treatment-emergent adverse events occurring in the six hours following administration of intravenous ibuprofen.
Time Frame: 6 hours
Population: This analysis was conducted on participants treated with a fever or pain indication that received only a single dose of intravenous ibuprofen
Measure: Number; unit: Number of Events
Groups:
- Fever: Intravenous ibuprofen (400 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 5-10 minute Treatment Period.
- Pain: Intravenous ibuprofen (800 mg intravenous ibuprofen administered intravenously over 5-10 minutes) will be administered as a single dose during the 5-10 minute Treatment Period.
Arm/Group | Fever | Pain
Number analyzed (Participants) | 1 | 96
Number of Events | 0 | 16

3. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting
Description: The change from baseline to one hour post administration of intravenous ibuprofen in vitals sign assessments (Temperature)
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Degree Fahrenheit
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
Degree Fahrenheit | -0.9 [-2.7 to 0.3] | -0.1 [-3.2 to 1.6]

4. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The change from baseline to one hour post administration of intravenous ibuprofen in vital sign assessments (Heart Rate).
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Beats Per Minute
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
Beats Per Minute | -2 [-16 to 8] | -1 [-34 to 62]

5. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The change from baseline to one hour post administration of intravenous ibuprofen in vital sign assessments (Respiratory Rate).
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: Breaths Per Minute
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
Breaths Per Minute | -1 [-5 to 2] | 0 [-17 to 14]

6. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The change from baseline to one hour post administration of intravenous ibuprofen in vital sign assessments (Systolic Blood Pressure).
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
mm Hg | -8 [-56 to 16] | -4 [-51 to 45]

7. Primary Outcome: To Determine the Safety of a Single Dose of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain in the Hospital Setting.
Description: The change from baseline to one hour post administration of intravenous ibuprofen in vital sign assessments (Diastolic Blood Pressure).
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Fever | Pain
Number analyzed (Participants) | 11 | 139
mm Hg | -4 [-16 to 4] | -3 [-49 to 41]

8. Secondary Outcome: To Determine the Efficacy of a Single Dose of 400 mg Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever
Description: The change in temperature from baseline over the 4 hours following intravenous ibuprofen administration
Time Frame: 4 hours
Measure: Mean (95% Confidence Interval); unit: Degree Fahrenheit
Arm/Group | Fever
Number analyzed (Participants) | 11
Degree Fahrenheit | -1.5 [-2.2 to -0.7]

9. Secondary Outcome: To Determine the Efficacy of a Single Dose of 800 mg Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Pain (Mild to Moderate or Moderate to Severe).
Description: The change in patient self-assessment of pain utilizing the visual analog scale (VAS) from baseline over the 4 hours following intravenous ibuprofen administration. The VAS is a continuous scale compromised of a horizontal line, one hundred millimeters in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between o and 100.
Time Frame: 4 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pain
Number analyzed (Participants) | 139
units on a scale | -27.1 [-33.5 to -20.7]

10. Secondary Outcome: To Determine the Safety of a Multiple Doses of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain
Description: The incidence of treatment-emergent serious adverse events occurring through extended dosing.
Time Frame: 24 hours
Measure: Number; unit: Number of Serious Adverse Events
Arm/Group | Fever | Pain
Number analyzed (Participants) | 10 | 43
Number of Serious Adverse Events | 0 | 1

11. Secondary Outcome: To Determine the Safety of a Multiple Doses of Intravenous Ibuprofen Administered Over 5-10 Minutes for the Treatment of Fever or Pain
Description: The incidence of treatment-emergent adverse events occurring through extended dosing.
Time Frame: 24 hours
Measure: Number; unit: Number of Events
Arm/Group | Fever | Pain
Number analyzed (Participants) | 10 | 43
Number of Events | 0 | 14

ADVERSE EVENTS:
Arm/Group | Fever | Pain
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/139
Other Adverse Events (participants affected / at risk) | 0/11 | 43/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fever (N=11) | Pain (N=139)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fever (N=11) | Pain (N=139)
Infusion Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 22 (24)
Infusion Site Warmth (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 8 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Breath Sounds Abnormal (Investigations) | 0 (0) | 4 (4)
Blood Creatinine Decreased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Dry Eyes (Eye disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Infusion Related Reaction (Immune system disorders) | 0 (0) | 1 (1)
Post Procedural Oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No